CLINICAL TRIAL: NCT03167541
Title: A Randomised, Single-dose, 2-way Crossover, Open-label, Comparative Bioavailability Study Comparing Test Naproxen Sodium Tablets (2 x 220 mg) With Commercially Available Reference Naproxen Sodium Tablets (2 x 220 mg) in the Fasted State
Brief Title: Naproxen Sodium (2 x 220 mg) Fasted Comparative Bioavailability Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Reckitt Benckiser Healthcare (UK) Limited (Industry)
Collaborators: Simbec Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: RB9-UK-1514
Record Dates: First submitted 2017-05-17; First posted 2017-05-30 (Actual); Results first posted 2019-02-28 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): Treatment Order: Test, Reference
  Interventions: Drug: Test; Drug: Reference
- 2 (Experimental): Treatment Order: Reference, Test
  Interventions: Drug: Test; Drug: Reference

INTERVENTIONS:
Drug: Test — RB naproxen sodium tablets (2x220mg)
Drug: Reference — Aleve naproxen sodium tablets (2x220mg)

SUMMARY:
This study is being conducted to investigate the rate and extent of naproxen absorption from the Test naproxen sodium formulation is bioequivalent to Aleve® naproxen sodium, a Reference product currently marketed in The Netherlands in order to support the registration of the Reckitt Benckiser (RB) naproxen sodium (220 mg tablets).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects who have given written informed consent.
2. Age: ≥ 18 years ≤ 50 years.
3. Body Mass Index (BMI) of ≥ 20 and ≤ 30 kg/m2.
4. Healthy as determined by past medical history, physical examination, vital signs, electrocardiogram (ECG), and laboratory tests at screening.
5. Female subject of child bearing potential with a negative pregnancy test at the screening visit and willing to use an effective method of contraception unless of non-childbearing potential or where abstaining from sexual intercourse in line with the preferred and usual lifestyle of the subject from first dose until 3 months after the final dose of study medication.
6. Female subject of non-child bearing potential with negative pregnancy test at the screening visit.
7. Male subject willing to use an effective method of contraception unless anatomically sterile or where abstaining from sexual intercourse in line with the preferred and usual lifestyle of the subject from first dose until 3 months after the final dose of study medication.

Exclusion Criteria:

1. Pregnant or lactating females.
2. Intention to become pregnant during the course of the study
3. Lack of safe contraception.
4. A history and/or presence of significant disease of any body system, including psychiatric disorders.
5. Any condition that may currently interfere with the absorption, distribution, metabolism or excretion of drugs.
6. A history of allergy or intolerance related to treatment with naproxen or other NSAIDs, or the excipients of the formulations.
7. A history of or active peptic or duodenal ulcers or gastro-intestinal bleed or upper gastro-intestinal bleed, or other significant gastro-intestinal disorders.
8. A history of frequent dyspepsia, e.g. heartburn or indigestion.
9. A history of migraine.
10. Current smokers and ex-smokers who have smoked or used nicotine replacement products during the previous 6 months prior to first dosing.
11. A history of substance abuse (including alcohol).
12. High consumption of stimulating drinks (coffee, tea, cola, energy drinks etc; total caffeine intake per day above 300 mg [1 cup of coffee equates to approximately 50 mg caffeine]).
13. Those with positive screen/test for drugs of abuse and alcohol.
14. Ingestion of a prescribed drug at any time in the 14 days before the first dose of study medication (excluding hormonal contraceptives and hormone replacement therapy), or consumption of enzyme inhibitors or inducers (drug, food or herb) 30 days prior to the first dose of study medication (such as barbiturates, carbamazepine, erythromycin, phenytoin, etc.).
15. Ingestion of an over-the-counter (OTC) preparation within 7 days before the first dose of study medication, including herbal medications, vitamin/fish oil supplements, naproxen and other NSAIDs.
16. Those who have consumed grapefruit or grapefruit juice, pummelo or Seville oranges in the 7 days prior to randomisation.
17. Strenuous physical exercise from 48 hours prior to randomisation to the post study Follow-Up Visit.
18. Donation of blood in quantity > 400 ml or other blood products e.g. to the blood transfusion service or significant loss of blood in the 12 weeks prior to screening.
19. Known human immunodeficiency virus (HIV) positive status, or a positive viral serology screen.
20. Topical use of naproxen within 7 days before the first dose of study medication.
21. Those previously randomised into this study.
22. Those who are an employee at the study site.
23. Those who are a partner or first degree relative of the Investigator.
24. Receipt of an investigational product, or participation in another trial involving a marketed or investigational drug in the 12 weeks prior to screening.
25. Those unable in the opinion of the Investigator to comply fully with the study requirements.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-10-12 (Actual); Primary Completion 2016-12-02 (Actual); Study Completion 2016-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Adams, MBBS, Principal Investigator — Simbec Research

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single-centre study conducted in United Kingdom.
Pre-assignment Details: Total 32 subjects were screened. Of these, 6 subjects were screen failures, 2 were surplus to requirement, 6 were reserve subjects. Subjects randomized were 18.
Groups:
- RB Naproxen (Test) First, Then Aleve Naproxen (Reference): Participants first received RB naproxen sodium 2 x 220 mg tablets single-oral dose in a fasting condition. After a washout period of 5-8 Days, they then received Aleve naproxen sodium 2 x 220 mg tablets single-oral dose in a fasting condition.
- Aleve Naproxen (Reference) First, Then RB Naproxen (Test): Participants first received Aleve naproxen sodium 2 x 220 mg tablets single-oral dose in a fasting condition. After a washout period of 5-8 Days, they then received RB naproxen sodium 2 x 220 mg tablets single-oral dose in a fasting condition.
Period: First Intervention
Arm/Group | RB Naproxen (Test) First, Then Aleve Naproxen (Reference) | Aleve Naproxen (Reference) First, Then RB Naproxen (Test)
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0
Period: Washout: 5-8 Days
Arm/Group | RB Naproxen (Test) First, Then Aleve Naproxen (Reference) | Aleve Naproxen (Reference) First, Then RB Naproxen (Test)
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | RB Naproxen (Test) First, Then Aleve Naproxen (Reference) | Aleve Naproxen (Reference) First, Then RB Naproxen (Test)
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: RB Naproxen Sodium 2 x 220 mg single dose by mouth under fasted condition.
  Aleve® Naproxen Sodium 2 x 220 mg single dose by mouth under fasted condition.
  There was a 5 to 8 days washout period between each administration.
Arm/Group | All Study Participants
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.6 (9.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 11
Race/Ethnicity, Customized [Number; unit: participants]
  White | 18
Height [Mean (Standard Deviation); unit: cm] | 172 (11.77)
Weight [Mean (Standard Deviation); unit: kg] | 74.69 (14.676)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 25.025 (2.7857)

OUTCOME MEASURES:

1. Primary Outcome: Area Under Plasma Concentration-time at Time t (AUC0-t)
Description: AUC0-t defines Area under the plasma concentration-time curve (AUC) from administration to the last quantifiable concentration at time t.
Time Frame: Pre-dose and at 15 mins, 30 mins, 45 mins, 1 hour, 1 hour 15 mins, 1 hour 30 mins, 1 hour 45 mins, 2 hours, 2 hours 30 mins, 3, 4, 6, 9, 15 (Day 1), 24, 36 (Day 2), 48 (Day 3) and 72 (Day 4) hours post-dose
Population: Pharmacokinetic (PK) Parameter Summary Set Population includes all subjects from the PK dataset with evaluable PK parameters for each treatment period.
Measure: Mean (Standard Deviation); unit: h*μg/mL
Groups:
- Test: RB Naproxen Sodium 2 x 220 mg: RB naproxen sodium 2 x 220 mg tablets single dose by mouth under fasted condition
- Reference: Aleve Naproxen Sodium 2x220 mg: Aleve naproxen sodium 2 x 220 mg tablets single dose by mouth under fasted condition.
Arm/Group | Test: RB Naproxen Sodium 2 x 220 mg | Reference: Aleve Naproxen Sodium 2x220 mg
Number analyzed (Participants) | 18 | 18
h*μg/mL | 915 (207) | 909 (186)

2. Primary Outcome: Maximum Plasma Concentration (Cmax)
Time Frame: as for outcome 1
Population: PK Parameter Summary Set Population
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Test: RB Naproxen Sodium 2 x 220 mg | Reference: Aleve Naproxen Sodium 2x220 mg
Number analyzed (Participants) | 18 | 18
μg/mL | 66.9 (11.9) | 65.2 (9.65)

3. Secondary Outcome: Elimination Rate Constant (Kel)
Description: Elimination Rate Constant (Kel) was calculated as the absolute value of the log-linear regression slope of the elimination phase (logged) over time (linear) using the post Cmax concentrations [at least 3 non-below the limit of quantification (BLQ)] that maximised the adjusted R2.
Time Frame: as for outcome 1
Population: PK Parameter Summary Set Population
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Test: RB Naproxen Sodium 2 x 220 mg | Reference: Aleve Naproxen Sodium 2x220 mg
Number analyzed (Participants) | 18 | 18
1/h | 0.0413 (0.00858) | 0.0414 (0.00673)

4. Secondary Outcome: Area Under the Plasma Concentration Curve From Administration to Infinity (AUC0-inf)
Description: Area under the plasma concentration curve from administration to infinity (AUC0-inf) was calculated as AUC0-t + (Ct/Kel) where Ct was the last quantifiable concentration at time t
Time Frame: as for outcome 1
Population: PK Parameter Summary Set Population
Measure: Mean (Standard Deviation); unit: h*μg/mL
Arm/Group | Test: RB Naproxen Sodium 2 x 220 mg | Reference: Aleve Naproxen Sodium 2x220 mg
Number analyzed (Participants) | 18 | 18
h*μg/mL | 972 (232) | 963 (203)

5. Secondary Outcome: Residual Area (AUC%Extrap)
Description: AUC%extrap represents the percentage of the AUC0-inf obtained by extrapolation, calculated as (1 - [AUC0-last/AUC0-inf]) multiplied by 100.
Time Frame: as for outcome 1
Population: PK Parameter Summary Set population
Measure: Mean (Standard Deviation); unit: Percentage of AUC
Arm/Group | Test: RB Naproxen Sodium 2 x 220 mg | Reference: Aleve Naproxen Sodium 2x220 mg
Number analyzed (Participants) | 18 | 18
Percentage of AUC | 5.68 (2.03) | 5.58 (1.72)

6. Secondary Outcome: Time Until Cmax is First Achieved (Tmax)
Time Frame: as for outcome 1
Population: PK Parameter Summary Set population
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Test: RB Naproxen Sodium 2 x 220 mg | Reference: Aleve Naproxen Sodium 2x220 mg
Number analyzed (Participants) | 18 | 18
hour | 1.38 (1.35) | 1.31 (1.28)

7. Secondary Outcome: Plasma Concentration (Elimination) Half-life (T1/2)
Time Frame: as for outcome 1
Population: PK Parameter Summary Set population
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Test: RB Naproxen Sodium 2 x 220 mg | Reference: Aleve Naproxen Sodium 2x220 mg
Number analyzed (Participants) | 18 | 18
hour | 17.3 (2.92) | 17.1 (2.48)

8. Secondary Outcome: Plasma Concentration at Each Planned Nominal Time-point (Cn)
Time Frame: as for outcome 1
Population: PK Parameter Summary Set population
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Test: RB Naproxen Sodium 2 x 220 mg | Reference: Aleve Naproxen Sodium 2x220 mg
Number analyzed (Participants) | 18 | 18
μg/mL
  Pre-dose | 0 (0) | 0 (0)
  15 mins | 15.6 (14.8) | 16.1 (12)
  30 mins | 49 (22.7) | 47.3 (23.3)
  45 mins | 58.4 (20) | 54.1 (22.4)
  1 hr | 57 (13.1) | 53.6 (18.7)
  1 hr 15 mins | 53.6 (10.4) | 52.9 (15.8)
  1 hr 30 mins | 55.9 (10.1) | 52.5 (14.2)
  1 hr 45 mins | 52.5 (8.54) | 54 (10.2)
  2 hrs | 51.4 (8.05) | 53.4 (9.13)
  2 hrs 30 mins | 48.3 (7.17) | 50 (8.47)
  3 hrs | 45 (6.34) | 47.1 (7.03)
  4 hrs | 40.8 (6) | 41.8 (6.36)
  6 hrs | 34.1 (6.34) | 34.6 (6.22)
  9 hrs | 6.34 (5.21) | 27.7 (5.25)
  15 hrs | 4.42 (23.5) | 18.9 (3.68)
  24 hrs | 3.61 (26.1) | 13.3 (3.08)
  36 hrs | 2.8 (35) | 7.9 (2.53)
  48 hrs | 1.98 (39) | 4.98 (1.89)
  72 hrs | 0.938 (42.3) | 2.15 (0.764)

9. Secondary Outcome: Occurrence of Adverse Events (AEs)
Description: Intensity was determined by the Investigator
  Mild = AE does not limit usual activities; subject may experience slight discomfort.
  Moderate = AE results in some limitation of usual activities; subject may experience significant discomfort.
  Severe = AE results in an inability to carry out usual activities; subject may experience intolerable discomfort or pain.
  Relationship to Investigational Medicinal Products (IMP)
  Certain = AE was definitely caused by IMP. Probable = Most likely that the AE was caused by IMP. Possible = Reasonable suspicion that the AE was caused by IMP Unlikely = Slight, but remote, chance that the AE was caused by IMP but the balance of judgment is that it was most likely not due to the IMP.
  Unrelated = No possibility that the AE was caused by IMP Un-assessable/Unclassified = Insufficient information to be able to make an assessment.
  Conditional/Unclassified = Insufficient information to make an assessment at present.
Time Frame: Up to follow-up day 7
Population: Safety population
Measure: Number; unit: Number of events
Groups:
- Reference: Aleve® Naproxen Sodium 2 x 220 mg: Aleve naproxen sodium 2 x 220 mg tablets single dose by mouth under fasted condition.
Arm/Group | Test: RB Naproxen Sodium 2 x 220 mg | Reference: Aleve® Naproxen Sodium 2 x 220 mg
Number analyzed (Participants) | 18 | 18
Number of events
  Treatment Emergent Adverse Event (TEAE) | 1 | 0
  Serious TEAE | 0 | 0
  TEAE Leading to Withdrawal | 0 | 0
  AE of mild intensity | 1 | 0
  AE of moderate intensity | 0 | 0
  AE of severe intensity | 0 | 0
  Certain related AE | 0 | 0
  Probable related AE | 0 | 0
  Possible related AE | 0 | 0
  Unlikely related AE | 1 | 0
  Unrelated related AE | 0 | 0
  Conditional/Unclassified related AE | 0 | 0
  Unassessable/Unclassifiable related AE | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to follow-up day 7
Description: Treatment-emergent adverse events (TEAEs), i.e., existing conditions that worsened or events that occurred during the course of the study after first administration of IMP and before the end of the study, are included.
Groups:
- Test: RB Naproxen Sodium 2 x 220 mg: RB Naproxen Sodium 2 x 220 mg single dose by mouth under fasted condition.
- Reference: Aleve® Naproxen Sodium 2 x 220 mg: Aleve Naproxen Sodium 2 x 220 mg single dose by mouth under fasted condition.
Arm/Group | Test: RB Naproxen Sodium 2 x 220 mg | Reference: Aleve® Naproxen Sodium 2 x 220 mg
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 1/18 | 0/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test: RB Naproxen Sodium 2 x 220 mg (N=18) | Reference: Aleve® Naproxen Sodium 2 x 220 mg (N=18)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No